CLINICAL TRIAL: NCT03525132
Title: Study of the Retinal Vascularization by Laser Doppler Velocimetry Coupled With an Adaptive Optics Camera ( AO-LDV) in Healthy Subject and Subject Affected by Glaucoma or Retinal Venous Occlusion
Brief Title: Study of the Retinal Vascularization by Laser Doppler Velocimetry Coupled With an Adaptive Optics Camera ( AO-LDV)
Acronym: AO-LDV
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2014-A01353-44
Record Dates: First submitted 2018-04-26; First posted 2018-05-15 (Actual); Last update posted 2019-06-17 (Actual); Status verified 2019-06

CONDITIONS: Glaucoma; Retinal Vein Occlusion
MeSH Terms: conditions — Glaucoma; Retinal Vein Occlusion | interventions — Laser-Doppler Flowmetry

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Healthy subjects (Experimental): 120 healthy subjects in the first session and 30 in the second Intervention : Laser Doppler Velocimetry + Optic Adaptative Camera
  Interventions: Procedure: Laser Doppler Velocimetry + Optic Adaptative Camera
- Glaucoma (Experimental): 60 subjects with glaucoma Intervention : Laser Doppler Velocimetry + Optic Adaptative Camera
  Interventions: Procedure: Laser Doppler Velocimetry + Optic Adaptative Camera
- Retinal vein occlusion (Experimental): 80 subjects with retinal vein occlusion including 40 with peripheric occlusion and 40 with central occlusion Intervention : Laser Doppler Velocimetry + Optic Adaptative Camera
  Interventions: Procedure: Laser Doppler Velocimetry + Optic Adaptative Camera

INTERVENTIONS:
Procedure: Laser Doppler Velocimetry + Optic Adaptative Camera — Fluxometry measure while subject is sitting in front of the optic adaptative camera

SUMMARY:
The difficulty to measure blood flow in humans is connected with the necessity of using not invasive, reliable and reproducible techniques.

There is several quantitative approaches to study eye blood flow which do not answer all these specifications. The laser doppler velocimetry allows movement speed measures but not vessel diameter. Optical coherence tomography doppler allows a simultaneous diameter and speed of travel (movement) measures, but presents a limited spatial resolution and thereby not easily reproducible vessel diameter measures.

The investigators propose development of a technique allowing a simultaneous diameter and velocity measure of these vessels.

DETAILED DESCRIPTION:
The eye blood flow plays a fundamental role in the eye physiology, insuring the metabolic contributions of various eye tissues, in particular those associated with the vision photochemical processes. Eye blood flow changes are involved in the physiopathology of several frequent eye diseases susceptible to lead to blindness (glaucoma,age-related macular degeneration, venous or arterial occlusions). Numerous systematic pathologies can also alter eye blood flow (diabetes, sleep apnea, arterial high blood pressure, inflammation).

The difficulty to measure blood flow in humans is connected with the necessity of using not invasive, reliable and reproducible techniques.

There is several quantitative approaches to study eye blood flow which do not answer all these specifications. The laser doppler velocimetry allows movement speed measures but not vessel diameter. Optical coherence tomography doppler allows a simultaneous diameter and speed of travel (movement) measures, but presents a limited spatial resolution and thereby not easily reproducible vessel diameter measures.

The investigators propose development of a technique allowing a simultaneous diameter and velocity measure of these vessels.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to give written Informed Consent and to comply with the requirements of the study protocol
* Person affiliated to social security
* Age between 18 and 80 years
* Capable of focusing a target without ocular micro stuttering
* For healthy subject : absence of ocular and systemic pathology and no medical treatment
* For subject with glaucoma : Primitive open-angle glaucoma unilateral or bilateral. Visual field must be considerate as compatible and reliable with campimetric impairment known in glaucoma.
* For subject wih retinal veinous occlusion : Retinal central vein occlusion or branch retinal vein occlusion medically confirmed with an eye fundus exam and fluorescein angiography.

Non-inclusion Criteria:

* Subject mentioned in L1121-5 to L1121-8 article of French Health Code : pregnant women, women capable of child bearing without contraceptive measures, under-age subject, subject under juridic protection or not able to give informed consent, subject deprived of liberty
* Any systemic medication with action on intraocular pressure such as sympathomimetic and beta blocker
* Hypersensitivity to tropicamide or its derivatives or to any eye drops excipients
* Subject who do not want to take part to the study
* Subject participating to another clinical trial
* Subject who can't come back for follow up visits
* Subject with lenses and who can't stop wearing them for the study protocol
* Close or narrow anterior chamber angle
* For healthy subject : Ametropia > 3 diopter, subject with non evolutive or evolutive ocular pathology
* For subject with glaucoma : Ametropia > 3 diopter, secondary glaucoma, closed angle glaucoma, isolated intraocular hypertonia, eye surgery within 3 months before the beginning of the study, trabeculoplasty, filtration surgery, associated evolutive or non-evolutive ocular pathology
* For subject with retinal veinous occlusion : Ametropia > 3, associated evolutive or non-evolutive ocular pathology, patient already treated with intravitreal injection with anti-VEGF or dexamethasone implant (no older than 4 months)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 290 (Estimated)
Dates: Start 2015-09-18 (Actual); Primary Completion 2020-03-18 (Estimated); Study Completion 2020-09-18 (Estimated)

PRIMARY OUTCOMES:
Change of total retinal blood flow in healthy subject | Day 0, Day 30 to Day 60
  Total retinal blood flow measurement in healthy subject at rest

SECONDARY OUTCOMES:
Repeatability and reproducibility of retinal blood flow measures intra and inter session | Day 0, Day 30 to Day 60
  Coefficient of variation for Repeatability and Reproducibility (3 measures session every 5 minutes on the same day, repeated one or two months after)
Change of retinal blood flow in different ages subjects | Day 0, Day 30 to Day 60
  Total retinal blood flow measurement in different ages subjects
Evaluation of the relation between retinal blood flow and vessel diameter | Day 0, Day 30 to Day 60
  Retinal blood flow and diameter of principal vessels coming from the optic disc
Measure retinal blood flow in subject with glaucoma and compare results with healthy subjects | Day 0
  Total retinal blood flow measured in subjects with glaucoma and age- and sex-matched healthy subjects
Measure retinal blood flow in subject with retinal vein occlusion and compare results with measurements made in ipsilateral non pathogenic vessels, controlateral vessels and healthy subjects. | Day 0, Month 1, Month 2, Month 3, Month 6
  Total blood flow compare to the controlateral eye and healthy subject data
Retinal blood flow evaluation after 1, 2 and 3 months after the inclusion of subject with retinal vein occlusion | Day 0, Month 1, Month 2, Month 3
  Partial retinal blood flow in a occluded temporal vein compare to a healthy ipsilateral temporal vein
Retinal blood flow evaluation after 1, 2, 3 and 6 months after intravitreal injection of aflibercept in subject treated for macular oedema as a complication of retinal vein occlusion | Day 0, Month 1, Month 2, Month 3, Month 6
  Retinal blood flow evolution will be evaluated regarding macular oedema and retinal ischaemia occurence

CONTACTS AND LOCATIONS:
Overall Officials: Florent Aptel, PhD, Principal Investigator — University Hospital, Grenoble
Locations (1):
- University Hospital Grenoble, Grenoble, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Evaluation du flux sanguin oculaire. In: Rapport SFO 2014 - Glaucome primitif à angle ouvert. — http://www.em-consulte.com/em/SFO/2014/html/file_100021.html